CLINICAL TRIAL: NCT02032381
Title: Prospective Study of Late Pulmonary Complications Occurring in Children Treated With Allogeneic Hematopoietic Stem Cells.
Brief Title: Prospective Study of Belated Pulmonary Complications Occurring in Children Treated With Allogeneic Hematopoietic Stem Cells.
Acronym: RESPPEDHEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P120137; 2013-A00966-39 (Other: APHP)
Record Dates: First submitted 2013-12-09; First posted 2014-01-10 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Bone Marrow Transplant Infection; Bronchiolitis Obliterans; Chronic Respiratory Insufficiency; Organizing Pneumonia; Pulmonary Cytolytic Thrombi
Keywords: non infectious pulmonary complications after hematopoietic cell transplant; functional respiratory test and exercise test; thoracic tomodensitometry
MeSH Terms: conditions — Bronchiolitis Obliterans; Organizing Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- allogeneic hematopoietic stem cell (Other): The eligible population for this study will consist of all children under 18 years who received allogeneic hematopoietic stem cell and evaluate of late pulmonary complications occurring in children treated with allogeneic hematopoietic stem cells.
  Interventions: Other: late pulmonary complications occurring in children treated with allogeneic hematopoietic stem cells.

INTERVENTIONS:
Other: late pulmonary complications occurring in children treated with allogeneic hematopoietic stem cells.

SUMMARY:
Hematopoietic stem cell transplantation (HSCT) is used to treat an expanding array of malignant and non-malignant disorders. This is a prospective multicenter study, in pediatric allo-BMT recipients to analyze the spectrum of noninfectious pulmonary complications (PC), to evaluate the prevalence and course of PFT abnormalities before and after transplant, and to detect risk factor for PC.

DETAILED DESCRIPTION:
It's a multicenter prospective study in France. All children under 18 years are included, just before the HSCT. The functional test before the HSCT at 6, 12, 18, 24, 30 and 36 months will be collected and a cardiopulmonary exercise test is done one and three years after the HSCT. Thoracic tomodensitometry is done before the HCT and after at 6, 12, 24 and 36 months.

All data will be collected upon the HSCT, the infections before and after the HSCT, the respiratory symptoms, and the treatment. Bronchia alveolar lavage and serum will be collected and frozen during the study.

The inclusion will be done during two years and children will be following during three years.

The purpose is to evaluate the prevalence, the course of PFT abnormalities before and after transplant, and to detect risk factor for PC.

ELIGIBILITY:
Inclusion Criteria:

* Age: from birth to 18 years
* Patient to be treated by allogeneic hematopoietic stem cell - Parents who have given their signed consent for the study
* Affiliation to a social security scheme

Exclusion Criteria:

* non exclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2014-01; Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Presence of belated non-infectious pulmonary complications | 3 years

SECONDARY OUTCOMES:
Presence of risk factors for belated non-infectious pulmonary complications | 3 years
Survival three years | 3 years
Severity of respiratory disease | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Houdouin Véronique, MD PHD, Principal Investigator — APHP
Locations (1):
- Houdouin véronique, Paris, France

REFERENCES:
- [Derived] Houdouin V, Feghali H, Boileau S, Guinot M, Reix P, Pages J, Crepon SG, Delclaux C. Prospective Evaluation of Cardiorespiratory Fitness After Hematopoietic Stem Cell Transplantation in Children. Pediatr Pulmonol. 2025 May;60(5):e70994. doi: 10.1002/ppul.70994. PMID 40371796
- [Derived] Houdouin V, Dubus JC, Crepon SG, Rialland F, Bruno B, Jubert C, Reix P, Pasquet M, Paillard C, Adjaoud D, Schweitzer C, Le Bourgeois M, Pages J, Yacoubi A, Dalle JH, Bergeron A, Delclaux C. Late-onset pulmonary complications following allogeneic hematopoietic cell transplantation in pediatric patients: a prospective multicenter study. Bone Marrow Transplant. 2024 Jun;59(6):858-866. doi: 10.1038/s41409-024-02258-7. Epub 2024 Mar 7. PMID 38454132